CLINICAL TRIAL: NCT01062503
Title: Duration of Suppression of Bone Turnover Following Treatment With Zoledronic Acid in Men With Metastatic Castration Resistant Prostate Cancer
Brief Title: Duration of Suppression of Bone Turnover Following Treatment With Zoledronic Acid in Men With Metastatic CRPC
Acronym: SubDueP
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB 09-0688-C; PRIT9 (Other Grant/Funding Number: Self); NCT01016171 (obsolete NCT alias)
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Prostate Cancer; Bone Metastasis
Keywords: Cancer; Prostate; metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Zoledronic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Zoledronic acid — ZA at a dose of 4mg will be administered by intravenous infusion over 15 minutes in at least 100mls of saline
  Other Names: Zometa

SUMMARY:
Bone is the most common site of metastases in prostate cancer and bone complications cause substantial morbidity to this population. Phase III studies have shown that zoledronic acid is effective in decreasing the morbidity associated with bone metastases. Zoledronic acid (ZA) is generally well tolerated but may have side effects such as hypocalcemia, renal impairment and osteonecrosis of the jaw. Administration of ZA as infrequently as once yearly is sufficient to prevent osteopenia or osteoporosis. The optimal treatment interval is unknown, but the drug is often empirically administered every 3-4 weeks. The cost of such treatment is high, and the risk of exposing patients (especially those at low risk) to potential serious side effects with uncertain benefit warrants investigation. This study will determine the duration of suppression of bone turnover in prostate cancer patients with bone metastases following a single infusion of Zoledronic Acid and its effect on quality of life.

DETAILED DESCRIPTION:
The bone is the most common site of metastasis in men with prostate cancer, and that bone metastases are associated with a significant risk of SREs. Prevention and delay in onset of SREs has been demonstrated with use of ZA. The optimal dosing frequency of ZA is not known in this population but it is usually given every 3-4 weeks, whereas injections as infrequently as once yearly protect from bone loss in patients without bone metastases who are receiving ADT. uNTX, sCTX and BAP are markers of bone turnover and bone formation that are suppressed in response to ZA and are associated with the likelihood of development of an SRE. In this study, we propose to determine the duration of suppression of bone turnover (all uNTX, sCTX and BAP) in response to a single dose of ZA in patients with castration resistant prostate cancer metastatic to bone.

Our objectives for this study:

1. To estimate the proportion of patients with suppression of bone turnover at 12 weeks after administration of a single dose of ZA.
2. To estimate the distribution of duration of suppression of bone turnover up to 12 weeks after administration of ZA.
3. To evaluate the frequency of SREs experienced by patients in this population.
4. To measure quality of life and presence of bone pain over a 12 week period in this patient population by utilizing the Functional Assessment of Cancer Therapy - Bone Pain (FACT-BP) and Brief Pain Inventory (BPI) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed prostate cancer that has become castration resistant
* Radiological or pathological evidence of bone metastases. (Positive bone scan, MRI, or CT or pathological fracture, or pathological sample from bone biopsy showing evidence of metastatic prostate cancer)
* Patient has not yet started on BP therapy for metastatic castration resistant prostate cancer
* Renal and hepatic function within the institutional normal range or at the discretion of the Investigator
* Age ≥ 18 years
* ECOG performance status ≤ 2
* Life expectancy >6 months
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Hypersensitivity or known allergy to bisphosphonates
* Patient who has received BP therapy for any reason within the past 1 year
* Acute or chronic renal insufficiency
* Evidence of infection/abscess on dental exam or recent dental extraction (within last 4 weeks)
* Acute pathological fracture, spinal cord compression, or hypercalcemia requiring urgent treatment (patient may enter study after acute issues are resolved)
* Patients with baseline hypocalcemia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a non-randomized observational study
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Patients given single dose of Zoledronic Acid 4mg IV | baseline

SECONDARY OUTCOMES:
Brief Pain Inventory Location Questionnaire | Baseline, Q6weeks, Q12weeks, 26weeks
FACT-BP Quality of Life Questionnaire | Baseline, Q6weeks, Q12weeks, 26weeks
We will monitor for uNTX, sCTX, BAP (fasting morning sample) | Baseline, Q3wks, Q6wks, Q9wks Q12wks

CONTACTS AND LOCATIONS:
Overall Officials: Ian F Tannock, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada